CLINICAL TRIAL: NCT05456971
Title: Evaluation of the Long Term Efficacy and Tolerability of ART FILLER® Volume and Lips, 2 Fillers Containing Hyaluronic Acid. Study ART FILLER 2
Brief Title: Evaluation of the Long Term Efficacy and Tolerability of ART FILLER® Volume and Lips
Acronym: AF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires FILLMED (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF2:2016-A00358-43
Record Dates: First submitted 2022-03-29; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Throughout the study period (18 months), only two products will be used for the aesthetic procedures (Art Filler® Volume and Art Filler® Lips). 100 subjects will be injected in order to have at least 100 midface regions and 100 lips treated and assessed at 3 or 6 weeks for the primary end point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art filler Volume (Experimental): To confirm the capacity of the VOLUME filler to restore a midface volume 3 weeks after the first injection or after 6 weeks if a touch up was performed at 3 weeks.
  Interventions: Device: Art Filler Volume
- Art Filler Lips (Experimental): To confirm the capacity of the LIPS filler to restored volume of the treated lip 3 weeks after the first injection or at 6 weeks if a top up at 3 weeks is performed.
  Interventions: Device: Art Filler Lips

INTERVENTIONS:
Device: Art Filler Volume — Midface correction with injectable hyaluronic acid based-filler
  Arms: Art filler Volume
Device: Art Filler Lips — Lipscorrection with injectable hyaluronic acid based-filler
  Arms: Art Filler Lips

SUMMARY:
The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume. These fillers (also known as soft tissue augmentation devices) can restore the age-related volume loss of the face, balance the disproportions or correct topographical anomalies. Art Filler® Volume and Art Filler Lips are two hyaluronic-based fillers. Both contain 0.3% lidocaine hydrochloride for its anaesthetic properties. The difference between the two devices lies in their viscosity, which must be adapted for the regions being treated and to restoring facial volumes. Midface for Art Filler® Volume and Lips for Art filler® Lips. On this background, a study is conducted to evaluate the long term efficacy and tolerability of Art Filler® Volume and Art Filler® Lips. It is a prospective, non-comparative, multicentre study with long term evaluation (18 months) of the tolerability and assessment of the efficacy of two devices containing hyaluronic acid intended for filling of lines and restoring volume to the face and lips.

DETAILED DESCRIPTION:
The function of injectable fillers for the treatment of dermal contour deformities is to smooth dermal depressions formed by the loss of volume. These fillers (also known as soft tissue augmentation devices) can restore the age-related volume loss of the face, balance the disproportions or correct topographical anomalies. Art Filler® Volume and Art Filler Lips are two hyaluronic-based fillers. Both contain 0.3% lidocaine hydrochloride for its anaesthetic properties. The difference between the two devices lies in their viscosity, which must be adapted for the regions being treated and to restoring facial volumes. Midface for Art Filler® Volume and Lips for Art filler® Lips. On this background, a study is conducted to evaluate the long term efficacy and tolerability of Art Filler® Volume and Art Filler® Lips. It is a prospective, non-comparative, multicentre study with long term evaluation (18 months) of the tolerability and assessment of the efficacy of two devices containing hyaluronic acid intended for filling of lines and restoring volume to the face and lips.

Primary objective:

* Art Filler® Volume: To confirm the capacity of Art Filler® Volume to restore a midface volume 3 weeks after the first injection or after 6 weeks if a touch-up was performed at 3 weeks. For a given target area (right or left) volume restoration will be deemed to be satisfactory if the Medicis Midface Volume Scale (MMVS) score falls by at least 1 moint compared to the baseline score.
* Art Filler® Lips: To confirm the capacity of Art Filler® Lips to restore volume of the treated lip 3 weeks after the first injection or after 6 weeks if a touch-up was performed at 3 weeks. For each lip treated (upper or lower) volume restoration will be deemed to be satisfactory if the Medicis Lip Fullness Scale (MLFS) score falls by at least 1 point compared to the baseline score.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects not under legal protection who have given their written agreement to take part.
2. Men or women, 19 years old or older with no upper limit.
3. Fitzpatrick phototype, I, II, III or IV.
4. Middle 1/3 of the face (cheeks/cheek pads): Score 3 or 4 (moderate to substantial loss of volume in the middle 1/3 of the face) on Medicis Midface Volume Scale (MMVS) AND/OR Lips: Score of 1 to 2 (very thin to thin lips) on the Medicis Lip Fullness Scale (MLFS)
5. Subjects seen at least 12 months after any aesthetic surgery procedure to the face.
6. Subjects at least 12 months from any corrective aesthetic facial injection (botulin in toxin or any filling agent) in the study regions, i.e. 1/3 of the midface and peri-oral/lip region.
7. Subjects who are members of a social security system.

Exclusion Criteria:

1. Subjects who do not meet the selection criteria.
2. Subjects participating in any other clinical study on the assessment of medicinal products or medical devices or subjects who are in the exclusion period following a clinical study.
3. Subjects who have received a facial injection/implantation of any non-resorbable filling agent.
4. Subjects with skin support devices (tension wires, gold wires or weave) in their face.
5. Subjects who have received laser or ultrasound medical treatment, deep chemical peeling or dermabrasion to the face during the previous 3 months or intending to undergo such a treatment to the face during the study.
6. Subjects with a known past history of hypertrophic, cheloid or dyschromic scarring.
7. Subjects with a past history of multiple severe allergies or anaphylactic shock.
8. Subjects with known hypersensitivity to any of the components of the study devices.
9. Subjects with porphyria.
10. Subjects with a past history of Streptococcal diseases (recurrent pharyngitis, acute articular rheumatic disease).
11. Subjects with hepatocellular impairment and coagulation disorders.
12. Subjects treated with medicinal products which reduce or inhibit liver metabolism.
13. Subjects with any acquired or congenital blood dyscrasia abnormality.
14. Subjects with cardiac conduction abnormalities.
15. Subjects with an episode of Herpes lesions on the face which have recovered within less than 4 weeks and with a contraindication to oral antiviral preventative treatment.
16. Subjects with facial scarring involving the injection regions.
17. Subjects receiving surgical orodental care and/or treatment for infection within 2 months.
18. Subjects receiving concomitant treatment (or treatment which has not been stopped for at least 3 months) with oral or injectable corticosteroids (inhaled corticosteroids and local corticosteroid therapy not involving the head or neck are permitted).
19. Subjects with concomitant treatment with an immunosuppressant or other chemotherapy treatment.
20. Subjects with a past history of radiotherapy to the head and neck within 6 months.
21. Subjects with a past history or autoimmune or connective tissue disease.
22. Subjects with an acute inflammatory reaction or bacterial or viral infection or seen within 1 month after the end of such an episode.
23. Pregnant or breast-feeding women (a urine pregnancy test will be performed before each injection).
24. Subjects suffering from epilepsy not controlled by treatment.
25. Subjects with a systemic or psychiatric disorder which could compromise their participation.
26. Receipt of an NSAID, or high dose vitamin C and/or E within one week.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Volume correction on D21 with Art Filler Volume | D21 (21 days after the injections)
  To confirm the capacity of Art Filler Volume to restore a midface volume 3 weeks (D21) after the first injection or after 6 weeks if a touch up was performed at 3 weeks. For a given target area (right or left) volume restoration will be deemed to be satisfactory if the MMVS (Medicis Midface Volume Scale) score falls by at least 1 point compared to the baseline score. (Score 1, Fairly full midface to Score 4, Substantial loss of fullness)
Volume correction on D21 with Art Filler Lips | D21 (21 days after the injections)
  To confirm the capacity of the LIPS filler to restored volume of the treated lip 3 weeks (D21) after the first injection or at 6 weeks if a touch up at 3 weeks is performed. For each lip treated (upper or lower), volume restoration will be deemed to be satisfactory if the MLFS (Medicis Lip Fullness Scale) increases by at least 1 point compared to the baseline score. (Score 1, very thin to Score 5, very full)..

SECONDARY OUTCOMES:
Description of local tolerability and emergent local and general incidents during a maximum follow up period of 18 months. | 18 months (540 Days after the injections)
  For each visit involving an injection, a descriptive analysis of immediate pain experienced (5 point verbal score completed for each target region treated) and effects detected will be performed. These events will be grouped according to the clinician's own wording, by type of event. They will also be categorised as local or systemic events. Their severity, persistence and causal relationship with the procedure will be described.
  An overall analysis will also be conducted including all injections administered over the 18 month follow up period. The prevalence of these events will be calculated taking account of the target area for local events.
Evaluation of persistence of volume-enhancing effect | 18 months (540 Days after the injections)
  The MMVS (Medicis Midface Volume Scale) and MFLS (Medicis Lip Fullness Scale) scores for each region injected measured at 3 weeks or at 6 weeks (if a top up is carried out at 3 weeks) after the first injection will define the optimal cosmetic score for a given target region.
Evaluation of overall cosmetic improvement | 18 months (540 Days after the injections)
  Overall cosmetic improvement will be reported for the PP (Per Protocol) population at 3/6 weeks and at 3, 6, 9, 12, 15 and 18 months from the Doctor and subject GAIS (Global Aesthetic Improvement Scale).
Evaluation of the injection procedures | 18 months (540 Days after the injections)
  Description of the procedures and injection volumes of the VOLUME filler and LIPS filler and the technical ease of use of these fillers at each visit involving an injection (for a given visit, the total volume injected will be the sum of the initial injection and any top up at 3 weeks). An overall descriptive analysis will also be conducted taking account of all of the injections administered over the whole follow up period.
Evaluation of self-esteem by subjects | 12 months (360 Days after the injections)
  The evaluation of self-esteem will be determined by using the ETES scale ( "Echelle toulousaine d'estime de soi"). The overall ETES score will be calculated at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ferial Fanian, MD, Study Director — Laboratoires FILLMED